CLINICAL TRIAL: NCT05060666
Title: Placebo-controlled Randomized Double-blind Phase III Study on the Efficacy and Safety of Ivermectin Tablets (Driponin®) for the Prophylaxis of COVID-19 Disease in Adult Contact Persons Living in the Household of a Person Suffering From COVID-19 [German: Placebo-kontrollierte Randomisierte Doppel-blinde Phase III Studie Zur Wirksamkeit Und Sicherheit Von Ivermectin Tabletten (Driponin®) für Die Prophylaxe Der COVID-19 Erkrankung Bei im Haushalt Lebenden Erwachsenen Kontaktpersonen Einer an COVID-19 Erkrankten Person]
Brief Title: Prophylaxis of COVID-19 Disease With Ivermectin in COVID-19 Contact Persons [German: Prophylaxe Der COVID-19-Erkrankung Mit Ivermectin Bei COVID-19 Kontaktpersonen]
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: GKM Gesellschaft für Therapieforschung mbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PREVENT-COVID; 2021-002445-15 (EudraCT Number)
Record Dates: First submitted 2021-09-28; First posted 2021-09-29 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: COVID-19 post-exposure prophylaxis
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin (Experimental): 2 doses of ivermectin at day 0 and day 2
  Interventions: Drug: Ivermectin
- Placebo (Placebo Comparator): 2 doses of placebo at day 0 and day 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin — 2 doses of Ivermectin will be administered with 48 hours time interval.
  The dosage is based on body weight calculated as follows:
  * 15 mg for 40-60 kg = 5 tablets à 3 mg
  * 18 mg for 60-80 kg = 6 tablets à 3 mg
  * 24 mg for > 80 kg = 8 tablets à 3 mg each
  This corresponds to an ivermectin dose of about 300 µg / kg.
  Other Names: Driponin; ATC-code P02CF01; Substance code SUB12089MIG
  Arms: Ivermectin
Drug: Placebo — An analogous number of tablets is administered for placebo:
  * 5 tablets for 40-60 kg
  * 6 tablets for 60-80 kg
  * 8 tablets for > 80 kg
  The size, appearance, smell and taste of the tablets of placebo are identical to Ivermectin.
  Arms: Placebo

SUMMARY:
The Prevent-COVID study is a prospective, multicenter, randomized, two-armed, placebo-controlled, double-blind, interventional study in which the efficacy and safety of ivermectin in COVID-19 post-exposure prophylaxis (PEP) is examined in adult, close family contacts living in the household of a subject suffering from COVID-19.

DETAILED DESCRIPTION:
Study population and study sites:

The study is carried out in about 30 private practices or clinics in Germany that regularly carry out SARS-CoV-2 PCR tests and treat COVID-19 patients.

Adult close contact persons of newly diagnosed COVID-19 patients living in the same household are considered for participation.

Study duration and assessment:

The study will last 14 days, in which the following study-specific measures will be undertaken:

* Documentation of demographics (age, gender, ethnicity, height and weight, degree of relationship to the COVID-19 patient)
* Documentation of current comorbidities
* Documentation of current medical accompanying measures
* Documentation of the general condition
* Vital signs
* COVID-19 symptoms
* SARS-CoV-2 PCR test: Only for medical confirmation of the presence of COVID-19 symptoms during an unplanned COVID-19 visit or final visit.
* Subject diary (daily measurement of body temperature, contact intensity with the index person)
* Pregnancy test in women of childbearing potential

Objectives:

Primary Objective: To demonstrate the efficacy of ivermectin in the COVID-19 post-exposure prophylaxis of adult contact persons living in the household of a person suffering from COVID-19 (index person)

Secondary objectives:

* To demonstrate the safety of ivermectin in the COVID-19 post-exposure prophylaxis of adult contact persons living in the household of a person suffering from COVID-19 (index person)
* To determine the severity of the symptoms of subjects suffering from COVID-19 during the study period and the comparison between the ivermectin and the placebo group.

IMP: Driponin® is an approved drug with the active ingredient Ivermectin, used to treat parasitic infections. One tablet Driponin® contains 3 mg Ivermectin. As part of the clinical trial, the medicinal product will be examined with regard to indication, dosage and application schedule deviating from the intended purpose and the package insert.

ELIGIBILITY:
Inclusion Criteria:

* age of at least 18 years
* adult subject living in the same household as a related COVID-19 patient (index person)

Exclusion Criteria:

* index person has COVID-19 symptoms for more than 5 days at enrolment
* known past COVID-19 or current infection confirmed by positive SARS-CoV-2 PCR test at enrolment
* symptoms at enrolment indicating COVID-19: increased body temperature OR acute respiratory symptoms of any severity OR newly occuring loss of taste or smell OR ague OR sumulatneously occuring headache and body ache
* known contraindications to the use of the study medication (in alignemnt with current summary of product characteristics of Driponin®)
* known chronic obstructive pulmonary disease
* known acute or chronic hepatitis B or C or other clinically recognizable or known liver dysfunction
* known HIV infection or AIDS
* known symptomatic allergic rhinitis
* current (inlcuding up to 24 hours before enrolment) or planned (during next 14 days) therapy with non-steroidal anti-inflammatory drugs, other pain medication (e.g., ASS (including prophylactic use), metamizol)
* recent (up to 28 days before enrolment) or planned (during next 14 days) therapy with systemic steroids
* recent (up to 28 days before enrolment) or planned (during next 14 days) therapy with systemic immunosuppressive drugs
* known or clinically suspected disturbance of the blood-brain-barrier (e.g., ABCB-1 (=MDR1) mutation) as well as history of neurotoxic effects by ivermectin or other substrates/inhibitors of the para-glycoprotein (P-gp)
* known hypersensitivity/intolerance to the study drug or any of its exicpients, in particular ivermectin, microcrystalline cellulose, pre-agglutinated starch, butyl hydroxyanisole or magnesium stearate
* pregnancy or lactation
* women of child-bearing potential planning to become pregnant or not using effective mehods of contraception
* any other severe disorder, which in the opinion of the investigator would preclude the subject from trial participation
* previous or planned (during next 14 days) vaccination with any COVID-19 vaccine
* recent (up to 28 days before enrolment) or planned (during next 14 days) therapy with Ivermectin
* recent (up to 28 days before enrolment) or planned (during next 14 days) therapy with drugs with evident or potential benefit in treating COVID-19 in alignemnt with RKI
* apparent unreliability or lack of compliance (e.g., not willing to orally administer the required number of tablets on 2 days or not willing to complete the subject diary during 14 days)
* known alcohol or drug abuse
* participation in another clinical trial during the last 30 days or planned participation in another clinical trial during the next 30 days
* previous participation in this same clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
COVID-19 disease | Day 14
  Occurrence of a COVID-19 disease up to the final visit (day 14), defined as the presence of the clinical condition according to the RKI case definition (acute respiratory symptoms of any severity OR new loss of smell and taste occurred OR illness-related death) AND a positive SARS-CoV-2 PCR test on the day the symptoms were determined (+/- 4 days)

SECONDARY OUTCOMES:
Adverse events and side effects | 14 days
  Number and severity of adverse events and side effects.
Type, number and severity of symptoms | 14 days
  Type, number and severity of symptoms within the 14-day of study on subjects suffering from COVID-19 (incl. hospitalization, oxygen saturation and demand, intensive care treatment)
Severity of the COVID-19 disease | 14 days
  Severity of the COVID-19 disease according to the investigator's assessment